CLINICAL TRIAL: NCT06110611
Title: Monolithic Zirconia Single Tooth Implant-supported Restorations With CAD/CAM Titanium Abutments in the Posterior Region: A 5-year Prospective Case Series Study
Brief Title: Monolithic Zirconia With CAD/CAM Titanium Abutments: A 5-year Prospective Case Series Study
Status: Enrolling by invitation | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, H.J.A. Meijer (Henny), Prof dr, University Medical Center Groningen
Other Study IDs: 18223
Record Dates: First submitted 2023-10-17; First posted 2023-10-31 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Edentulous Alveolar Ridge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- dental implant and a screw-retained implant-supported zirconia restoration: patients which were treated 5 years ago with a dental implant and a screw-retained implant-supported zirconia restoration
  Interventions: Device: Astra Tech Osseospeed EV® dental implant

INTERVENTIONS:
Device: Astra Tech Osseospeed EV® dental implant — Prospective study of a group of 50 patients which were treated 5 years ago with a dental implant and a screw-retained implant-supported zirconia restoration because of a missing tooth in the posterior region.
  Other Names: Atlantis™ CustomBase abutment with full-contour zirconia Atlantis® Crown

SUMMARY:
* Background There is a growing interest in restoring function in the posterior maxilla and mandible with dental implants. Next to this, these implants must be restored with crowns which are subject to minimal complications. Companies have introduced the option of screw-retaining and zirconia as crown material. The combination of posterior implants and screw-retained zirconia crowns are widely used, but prospective research on clinical performance and patient centered outcomes are scarce. Even more, 5-years data are lacking.
* Main research question To evaluate the clinical performance of Astra Tech Implants EV and Atlantis CustomBase Abutments with full-contour zirconia Atlantis Crowns in the posterior maxilla and mandible. The primary objective of the study is marginal bone level changes by radiological assessments at 5-years follow-up. Secondary objectives are implant and restoration survival, condition of peri- implant mucosa and patients' satisfaction.
* Design (including population, confounders/outcomes) The study design is an observational study of a group of patients which were treated 5 years ago with a dental implant and a screw-retained implant-supported zirconia restoration because of a missing tooth in the posterior region. Outcomes: primary outcome is the change in marginal peri-implant bone level 5 years after placing the definitive restoration. Secondary outcome measures will be implant and restoration survival, peri-implant mucosa health and patients' satisfaction using a questionnaire.

DETAILED DESCRIPTION:
• Introduction and rationale Nowadays, the use of dental implants for oral rehabilitation is a generally accepted treatment modality. During the first years of implant dentistry, dental implants were used mainly for the restoration of edentulous mandibles with implant-supported prostheses. Yet, there is a shift towards the application of dental implants for single-tooth replacements, supported by long-term studies reporting excellent survival rates. Not only in the aesthetic region, but also in the posterior maxilla and mandible there is a growing interest in restoring function. Dental implants show a good performance in the posterior region; in recent years attention has been shifted towards a better initial stability to reduce treatment time. Next to this, implants must be restored with crowns which are subject to minimal complications. Specially for the posterior region, companies have introduced the option of screw-retaining and zirconia as crown material, of which less technical complications are mentioned. The combination of posterior implants and screw-retained zirconia crowns are widely used, but prospective research on clinical performance and patient centered outcomes are scarce and 5-years results are lacking.

RESEARCH QUESTION To evaluate the clinical performance of Astra Tech Implants EV and Atlantis CustomBase Abutments with full-contour zirconia Atlantis Crowns in the posterior maxilla and mandible after a 5-years follow-up.

STUDY DESIGN The study design is an observational study of a group of 50 patients which were treated 5 years ago with a dental implant and a screw-retained implant-supported zirconia restoration because of a missing tooth in the posterior region.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the department of Oral and Maxillofacial Surgery 5 years ago and treated with a dental implant and a screw-retained implant-supported zirconia restoration because of having a missing tooth in the posterior region. At the time of treatment:
* The patient was 18 years or older;
* The missing tooth was a premolar or molar in maxilla or mandible;
* Sufficient healthy and vital bone to insert a dental implant with a minimum length of 8 mm and at least 4.2 mm in diameter with initial stability > 45 Ncm
* The implant site was free from infection;
* Adequate oral hygiene (modified plaque index and modified sulcus bleeding index ≤ 1);
* Sufficient mesio-distal, bucco-lingual, and interocclusal space for placement of an anatomic restoration;
* The patient was capable of understanding and giving informed consent.

Exclusion Criteria:

* Medical and general contraindications for the surgical procedures;
* Presence of an active and uncontrolled periodontal disease;
* Bruxism;
* Smoking
* A history of local radiotherapy to the head and neck region.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population: Patients referred to the department of Oral and Maxillofacial Surgery 5 years ago and treated with a dental implant and a screw-retained implant-supported zirconia restoration because of having a missing tooth in the posterior region. At the time of treatment:
  * The patient was 18 years or older;
  * The missing tooth was a premolar or molar in maxilla or mandible;
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in peri-implant marginal bone level (in millimetres) | 5 years
  Difference in peri-implant bone level measured in millimetres

SECONDARY OUTCOMES:
Implant survival and restoration survival (in percentage) | 5 years
  Percentage of initially placed implants and restorations still in place after 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Henny Meijer, prof dr, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No